CLINICAL TRIAL: NCT01775787
Title: Effects of Electronic Cigarettes on Nicotine Concentrations Before and 5, 10, 15, 20 and 30 Minutes After Use
Brief Title: Effects of Electronic Cigarettes on Nicotine Concentrations
Acronym: ECIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Cheryl Oncken, Professor, Department of Medicine, UConn Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ECIG 13-002-3
Record Dates: First submitted 2012-10-12; First posted 2013-01-25 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-10

CONDITIONS: Health Behavior
Keywords: smoking
MeSH Terms: conditions — Health Behavior; Smoking | interventions — Nicotine; Tobacco Products; Menthol; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tobacco Flavor/ Tobacco & Menthol Flavor (Other): Subjects randomized to Tobacco Flavor group 7-10 days, then crossed over to Tobacco and Menthol Flavor for 7-10 days.
  Nicotine with Tobacco Flavor and Tobacco & Menthol Flavor (18mg/mL nicotine)
  Interventions: Drug: Nicotine with Tobacco Flavor and Tobacco & Menthol Flavor
- Tobacco & Menthol Flavor/Tobacco Flavor (Other): Subjects randomized to Tobacco and Menthol Flavor for 7-10 days,then crossed over to Tobacco Flavor for 7-10 days.
  Nicotine with Tobacco Flavor and Tobacco & Menthol Flavor (18mg/mL nicotine)
  Interventions: Drug: Nicotine with Tobacco Flavor and Tobacco & Menthol Flavor

INTERVENTIONS:
Drug: Nicotine with Tobacco Flavor and Tobacco & Menthol Flavor — Subjects randomized to either Tobacco Flavor group for 7-10 days than crossed over to Tobacco & Menthol Flavor for 7-10 days or Tobacco & Menthol Flavor group for 7-10 days than crossed over to Tobacco Flavor for 7-10 days
  Other Names: Tobacco Flavor; Tobacco & Menthol Flavor; Electronic Cigarette; Nicotine

SUMMARY:
This study will examine whether nicotine levels increase with electronic cigarettes. It will also examine whether electronic cigarettes alter lung function tests. The study will obtain preliminary data on the medical effects of electronic cigarettes, with two different nicotine flavors, tobacco and tobacco with menthol, which are available for over the counter purchase.

The electronic cigarettes and juice used in this study is available for purchase through the internet. An investigational new drug application (IND) is not needed for this study.

DETAILED DESCRIPTION:
This is a randomized two-period cross-over study in which subjects who smoke greater than 10 cigarettes will be instructed to quit smoking and use either Joye (Ego C brand) with an 18 mg cartridge containing either a tobacco or tobacco mentholated flavor for one week. Prior to starting e-cig use we will collect one blood sample for nicotine/cotinine as a measure of overall nicotine exposure. Subjects will use the device for one week and at the end of approximately one week of use, we will assess nicotine/cotinine concentrations (before and 5, 10, 15, 20 and 30 minutes after the onset of ECIG use), pulmonary function tests (before and 5 minutes after ECIG use), and subjective impressions of satisfaction. At the end of one week, subjects will be crossed over to the other condition and assessments will be repeated after another week of E-cigarette use.

A total of 30 smokers will be recruited from the surrounding areas via advertisements in newspapers and radio advertisements and University of Connecticut Health Center (UCHC) broadcast e-mail. Posters will be placed in clinical areas to recruit from physician practices. Current smokers are being proposed for three reasons: 1) we wish to determine whether nicotine levels from e-cigarettes rise to the levels of regular cigarettes when used by regular smokers; 2) we wish to determine if there are any differences seen in pulmonary function when a person switches from regular cigarettes to e-cigarettes; 3) we wish to evaluate the level of satisfaction that regular smokers have with e-cigarettes. All of these questions will have implications for later, more extensive studies of e-cigarettes, particularly in regard to their utility as a smoking cessation modality.

Once a potential study subject calls and expresses interest in the study, preliminary inclusion criteria will be assessed over the phone. Inclusion criteria include 1) at least 18 years of age; 2) current use of at least 10 cigarettes daily; 3) willing to abstain from cigarette smoking, and substitute e-cigs, for approximately 2 weeks; 4) able to read and sign a consent form; Exclusion criteria: 1) unstable medical or psychiatric disorders as determined by the principal investigator; 2) pregnancy; 3) known hypersensitivity to nicotine or propylene glycol or menthol; 4) previous myocardial infarction (M.I.) or stroke; 5) uncontrolled hypertension [Blood pressure (BP) >160/100); 6) insulin dependent diabetes; 7) known chronic obstructive pulmonary disease (COPD) or asthma.

ELIGIBILITY:
Inclusion Criteria:

* Smoking 10 cigarettes daily
* Agree to abstain from smoking and use electronic cigarettes for 2 weeks

Exclusion Criteria:

* Unstable medical or psychiatric disorders as determined by the principal investigator
* Pregnancy
* Known hypersensitivity to nicotine or propylene glycol or menthol
* Recent M. I. or stroke
* Uncontrolled hypertension (BP.>160/100)
* Insulin dependent diabetes
* Known COPD or asthma
* Alcohol or other drug abuse or dependence

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Oncken, M.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oncken CA, Litt MD, McLaughlin LD, Burki NA. Nicotine concentrations with electronic cigarette use: effects of sex and flavor. Nicotine Tob Res. 2015 Apr;17(4):473-8. doi: 10.1093/ntr/ntu232. PMID 25762758
- See also: Nicotine concentrations with electronic cigarette use: effects of sex and flavor — https://www.ncbi.nlm.nih.gov/pubmed/25762758

RESULTS

PARTICIPANT FLOW:
Groups:
- Tobacco Flavor/ Tobacco & Menthol Flavor: Subjects randomized to Tobacco Flavor group 7-10 days, then crossed over to Tobacco and Menthol Flavor for 7-10 days.
  Nicotine with Tobacco Flavor or Tobacco & Menthol Flavor (18mg/mL nicotine
- Tobacco & Menthol Flavor/Tobacco Flavor: Subjects randomized to Tobacco and Menthol Flavor for 7-10 days,then crossed over to Tobacco Flavor for 7-10 days.
  Nicotine with Tobacco Flavor or Tobacco & Menthol Flavor (18mg/mL nicotine)
Period: First 7-10 Days
Arm/Group | Tobacco Flavor/ Tobacco & Menthol Flavor | Tobacco & Menthol Flavor/Tobacco Flavor
Started | 13 | 14
Completed | 12 | 8
Not Completed | 1 | 6
Not completed — Adverse Event | 0 | 1
Not completed — family emergency | 0 | 1
Not completed — time commitment | 0 | 2
Not completed — concerns with using IV | 1 | 2
Period: Second 7-10 Days
Arm/Group | Tobacco Flavor/ Tobacco & Menthol Flavor | Tobacco & Menthol Flavor/Tobacco Flavor
Started | 12 | 8
Completed | 12 | 6
Not Completed | 0 | 2
Not completed — time commitment | 0 | 1
Not completed — concerns with using IV | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis Nicotine Concentrations before ad 5 minutes after Ecig use, regardless of flavor.
Groups:
- Nicotine With Tobacco Flavor and With Tobacco & Menthol Flavor: Smokers were assigned to electronic cigarettes containing 18mg/mL of nicotine in either a tobacco flavor solution or a tobacco and menthol flavor solution and then switched to other flavor for an additional 7 to 10 days. Monitoring sessions occurred on the last day of trial period of each flavor.
Arm/Group | Nicotine With Tobacco Flavor and With Tobacco & Menthol Flavor
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Effects E-cig Use on Venous Nicotine Concentrations Before and 5 Minutes After Use
Description: To determine the effects of acute E-cig use on venous nicotine concentrations 5 minutes before and 5 minutes after 7-10 days of e-cigarette use.
Time Frame: 7-10 days
Population: Nicotine Concentrations Before and 5 Minutes After Ecig Use were intended to be analyzed, regardless of flavor, as pre-specified in the study protocol,
Measure: Mean (Standard Error); unit: ng/ml
Groups:
- Tobacco Flavor: Subjects received tobacco flavored nicotine for 7-10 days
- Tobacco & Menthol Flavor: Subjects received tobacco & menthol flavored nicotine for 7-10 days
Arm/Group | Tobacco Flavor | Tobacco & Menthol Flavor
Number analyzed (Participants) | 20 | 18
ng/ml
  Before Ecig used | 4.30 (.66) | 4.11 (1.23)
  5 minutes after ecig use | 8.66 (.08) | 8.77 (1.53)

ADVERSE EVENTS:
Time Frame: Period from Randomization to close of study
Groups:
- Tobacco Flavor & Tobacco & Menthol Flavor (TOB Flavor): AE occurred in intervention "Tobacco Flavor Session 17-10 days"
  Subjects randomized to Tobacco Flavor group 7-10 days, then crossed over to Tobacco and Menthol Flavor for 7-10 days.
  Nicotine with Tobacco Flavor or Tobacco & Menthol Flavor (18mg/mL nicotine)
- Tobacco Flavor & Tobacco & Menthol Flavor (TOB/MENTH Flavor): AE occurred in intervention "Tobacco Flavor Session 27-10 days"
  Subjects randomized to Tobacco Flavor group 7-10 days, then crossed over to Tobacco and Menthol Flavor for 7-10 days.
  Nicotine with Tobacco Flavor or Tobacco & Menthol Flavor (18mg/mL nicotine)
- Tobacco & Menthol Flavor & Tobacco Flavor (TOB/MENTH Flavor): AE occurred in intervention "Tobacco & Menthol Flavor Session 17-10 days"
  Subjects randomized to Tobacco & Menthol Flavor group 7-10 days, then crossed over to Tobacco Flavor for 7-10 days.
  Nicotine with Tobacco Flavor or Tobacco & Menthol Flavor (18mg/mL nicotine)
- Tobacco & Menthol Flavor & Tobacco Flavor (TOB Flavor): AE occurred in intervention "Tobacco Flavor Session 2 7-10 days"
  Subjects randomized to Tobacco & Menthol Flavor group 7-10 days, then crossed over to Tobacco Flavor for 7-10 days.
  Nicotine with Tobacco Flavor or Tobacco & Menthol Flavor (18mg/mL nicotine)
Arm/Group | Tobacco Flavor & Tobacco & Menthol Flavor (TOB Flavor) | Tobacco Flavor & Tobacco & Menthol Flavor (TOB/MENTH Flavor) | Tobacco & Menthol Flavor & Tobacco Flavor (TOB/MENTH Flavor) | Tobacco & Menthol Flavor & Tobacco Flavor (TOB Flavor)
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/14 | 0/8
Other Adverse Events (participants affected / at risk) | 1/13 | 0/12 | 6/14 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tobacco Flavor & Tobacco & Menthol Flavor (TOB Flavor) (N=13) | Tobacco Flavor & Tobacco & Menthol Flavor (TOB/MENTH Flavor) (N=12) | Tobacco & Menthol Flavor & Tobacco Flavor (TOB/MENTH Flavor) (N=14) | Tobacco & Menthol Flavor & Tobacco Flavor (TOB Flavor) (N=8)
Thoat itchy and cough (General disorders) | 0 | 0 | 1 | 0 — HEENT ( head, ears, eyes, nose and throat)
Concerns with using IV (Product Issues) | 0 | 0 | 2 | 1
Time Commitment (Social circumstances) | 0 | 0 | 2 | 1
Family Emergency (Social circumstances) | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes